CLINICAL TRIAL: NCT01825694
Title: An Integrated Treatment for Comorbid PTSD and Substance Abuse in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA031301 (NIH)
Record Dates: First submitted 2012-07-18; First posted 2013-04-08 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Substance Abuse; Traumatic Stress
Keywords: Substance Abuse; Traumatic Stress
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): The Standard of Care condition includes: 1) an individual session with the counselor, once per week; 2) a treatment group with the counselor, twice per week; and 3) parents of youth are invited to attend parent-only educational sessions weekly.
- Trauma-focused Substance Abuse Intervention (Experimental): See Intervention Arm description.
  Interventions: Behavioral: Trauma-focused Substance Abuse Intervention

INTERVENTIONS:
Behavioral: Trauma-focused Substance Abuse Intervention — An integrated treatment approach to reduce substance use and PTSD symptoms. The intervention program includes: 1) 1-2 individual sessions during which youth talk about the trauma, during the course of the intervention program; 2) 16 group sessions for youth; 3) 2 conjoint sessions with parents to improve communication and problem-solving skills; and 4) 2 parent-education group sessions.
  Arms: Trauma-focused Substance Abuse Intervention

SUMMARY:
This study plans to develop an integrated treatment for comorbid post-traumatic stress disorder (PTSD) and substance abuse (SA) in adolescents. The investigators aim to develop a treatment approach that is community-friendly, well-tolerated, and deliverable by substance abuse counselors (SAC) in outpatient settings. The proposed Trauma-Focused Substance Abuse Treatment (TFSAT) aims to reduce PTSD symptoms and substance use and build coping skills. The investigators propose to adapt an evidence-based trauma program, Cognitive-Behavioral Intervention for Trauma in Schools (CBITS), for adolescent substance abusers (ASAbusers); to assess the acceptability and feasibility of the integrated approach; and to pilot test the new program against standard care.

The investigators hypothesize that the intervention group, compared to the control group, will reduce substance use and symptoms for traumatic stress.

ELIGIBILITY:
Inclusion Criteria: Youth

* Between ages of 13 & 19;
* meeting DSM IV criteria for substance abuse/dependence and PTSD;
* previously enrolled at recruitment site for at least 2 weeks;
* parent/guardian provides permission for minors to participate.

Exclusion Criteria: Youth

* Not within the specified age range;
* presence of organic brain damage;
* inability to understand enrollment forms (e.g. Informed Assent/Consent Form)

Inclusion Criteria: Parents/Guardians

* Age 18 or above;
* parents/guardians of youth who meets inclusion criteria.

Exclusion Criteria: Parents/Guardians

* presence of organic brain damage.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-back (TFLB) Assessment of Substance Use | Participants will be followed for an expected average of 12 weeks.
  The TLFB uses a blank calendar form and a series of questions to cue recall of alcohol and drug (AOD) use. The investigators will use the TLFB interview technique to assess AOD use weekly.
Urine Toxicology Screen (UTS) | Participants will be followed for an expected average of 12 weeks.
  Urine samples will be collected twice per week at the treatment site to ensure validity of self-reports.
Child PTSD Symptom Scale (CPSS) | Change from Baseline in Child PTSD Symptom Scale at 8 weeks and change from Baseline in Child PTSD Symptom Scale at 12 weeks.
  The CPSS will assess for severity of traumatic stress symptoms.

SECONDARY OUTCOMES:
Child Post-Trauma Attitudes Scale (C-PTAS) | Baseline & 8 weeks & 3 months
  The C-PTAS will be used to assess trauma-related attitudes and beliefs.
Strengths & Difficulties Questionnaire (SDQ) | Baseline & 8 weeks & 3 months
  The SDQ will be used to assess parent-report of behavioral problems.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy S Wu, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Behavioral Health Services, Los Angeles, California, United States